CLINICAL TRIAL: NCT04362683
Title: Loop Recorder Evaluation in Patients Treated With High Power Short Duration Ablation for Paroxysmal Atrial Fibrillation With High Density Multi Directional Mapping (LOWE AF HD Study)
Brief Title: High Power Short Duration Ablation for Paroxysmal AF With High Density Multi Directional Mapping (LOWE AF HD Study).
Acronym: LOWE-AF-HD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gregorio Covino (Other)
Responsible Party: Sponsor-Investigator, Gregorio Covino, Principal Investigator, Ospedale S. Giovanni Bosco
Organization: Ospedale S. Giovanni Bosco (Other)
Other Study IDs: SGB01
Record Dates: First submitted 2020-04-07; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Atrial Fibrillation
Keywords: AF; High Power - Short Duration Ablation; High Density Mapping
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High Power Atrial Fibrillation Ablation: In our center, routine medical care for atrial fibrillation ablation includes:
  * Multidirectional high-density mapping
  * High power - short duration settings
  * Contact force sensing ablation catheter

SUMMARY:
The LOWE AF HD is a prospective, single-center, non-randomized study to assess safety, efficacy, acute and long-term outcome data of a specific ablation approach as treatment of paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
Pulmonary vein isolation using radiofrequency (RF) ablation is acknowledged used treatment strategy for atrial fibrillation, many different approaches are recently implemented. The specific approach used in this study includes:

* Multi-directional high-density mapping
* High power - short duration settings
* Contact force sensing ablation catheter The aim of LOWE AF HD is to assess the acute safety and success rate of this approach and also the long-term outcome assessed by atrial recurrences arrythmias collected by an implantable loop recorder.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive and unselected patients with a class I-IIa indication for ablation of paroxysmal AF
* 18 Years and older.
* Able and willing to provide written informed consent prior to any clinical investigation related procedure
* Able and willing to complete all required study procedures through 12 months
* Life expectancy less than 12 months

Exclusion Criteria:

* Persistent or long-standing persistent AF
* Presence of thrombus in left atrium and left atrium appendage
* MI, CABG or PCI within preceding 3 months
* Left atrial diameter > 5.0 cm
* LVEF < 35%
* NYHA class III or IV
* Previous atrial fibrillation ablation procedure with high density and high-power short duration approach
* Previous tricuspid or mitral valve repair surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for participation in the study have indication for ablation of paroxysmal AF and are eligible for PVI by catheter ablation based on the respective ACC/AHA/ESC Guideline valid at the date of procedure.
Sampling Method: Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2020-04-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Acute Procedural Success Rate | 1 day
  Acute procedural success defined as electrical isolation of all pulmonary veins, confirmed by the high-density voltage remap and loss of pace capture along ablation line after complete isolation.
Rate of patients without Atrial Fibrillation recurrences | 12 months after 3-months blanking period
  Freedom from Atrial Fibrillation (AF) defined as any documented recurrence of AF and/or atrial tachycardia (AT) and /or atrial flutter (AFL), lasting longer than 30 second, assessed from the end of the 3-months blanking period to 12 months following a single ablation procedure and collected by Implantable Loop Recorder (ILR).

SECONDARY OUTCOMES:
Adverse events rate | 1 month
  Procedural and post procedural safety assessed by reporting all adverse events in the first 30 days after ablation
Ablation Procedure Time | 1 day
  Complete procedure time (minutes)
Ablation Fluoroscopic Time | 1 day
  Fluoroscopic time recorded (minutes) during ablation procedure
Number of radiofrequency applications | 1 day
  Number of radiofrequency applications reported for each patient during ablation procedure.
Total radiofrequency ablation time | 1 day
  Total time (minutes) of radiofrequency applications in each patient during ablation procedure.
First pass pulmonary vein isolation | 1 day
  Number of patients in which PV isolation is obtained at first attempt.
Number of atrial fibrillation events | 12 months
  Number of AF events symptomatic and asymptomatic assessed from the end of the 3-months blanking period to 12 months following a single ablation procedure and collected by Implantable Loop Recorder (ILR).
Atrial Fibrillation Burden | 12 months
  AF Burden (in minutes) recorded at 12 months (after 3-months blanking period) of follow-up by Implantable Loop Recorder.

CONTACTS AND LOCATIONS:
Overall Officials: Gregorio Covino, MD, Principal Investigator — Ospedale San Giovanni Bosco
Locations (1):
- Ospedale San Giovanni Bosco, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Undecided